CLINICAL TRIAL: NCT00284817
Title: Phase I Study of MEDI522, a Humanized Monoclonal Antibody Directed Against the Human Alpha V Beta 3 Integrin, in Patients With Irinotecan-Refractory Advanced Colorectal Cancer or Other Solid Tumors Refractory to Standard Therapy
Brief Title: Phase I Study of MEDI522 in Patients With Irinotecan-Refractory Advanced Colorectal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Luz Hammershaimb, M.D., V.P., Clinical Dev., MedImmune LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MI-CP068
Record Dates: First submitted 2006-01-31; First posted 2006-02-01 (Estimated); Last update posted 2008-05-29 (Estimated); Status verified 2008-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — etaracizumab

ARMS (5):
- 1 (Experimental): MEDI-522
  Interventions: Drug: MEDI-522
- 2 (Experimental): MEDI-522
  Interventions: Drug: MEDI-522
- 3 (Experimental): MEDI-522
  Interventions: Drug: MEDI-522
- 4 (Experimental): MEDI-522
  Interventions: Drug: MEDI-522
- 5 (Experimental): MEDI-522
  Interventions: Drug: MEDI-522

INTERVENTIONS:
Drug: MEDI-522 — Administered as a 30-minute IV infusion; 4 mg/kg on Study Day 0 followed by weekly maintenance doses of 1 mg/kg for 51 weeks.
  Arms: 1
Drug: MEDI-522 — Administered as a 30-minute IV infusion; 4 mg/kg on Study Day 0 followed by weekly maintenance doses of 2mg/kg for 51 weeks.
  Arms: 2
Drug: MEDI-522 — Administered as a 30-minute IV infusion; 6 mg/kg on Study Day 0 followed by weekly maintenance doses of 2mg/kg for 51 weeks.
  Arms: 3
Drug: MEDI-522 — Administered as a 30-minute IV infusion; on Study Day 0 followed by weekly maintenance doses of 3mg/kg for 51 weeks.
  Arms: 4
Drug: MEDI-522 — The next cohort of patients will be treated after at least 3 of 4 patients treated in the previous cohort receive at least 3 weeks of treatment and experience no dose-limiting toxicity (DLT).
  Arms: 5

SUMMARY:
- Assess the safety and tolerance of a weekly MEDI522 regimen in patients with irinotecan-refractory advanced CRC or other solid tumors refractory to standard therapy.

DETAILED DESCRIPTION:
* Assess the safety and tolerance of a weekly MEDI 522 regimen in patients with irinotecan-refractory advanced CRC.
* Determine a Phase II recommended dose based on acceptable dose-limiting toxicity. Other considerations such as pharmacokinetic parameters may also be factored into the determination of a Phase II dose.

The secondary objectives of the study are to:

* Assess any antitumor activity of MEDI-522 in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed advanced CRC that has progressed through an irinotecan-containing regimen for metastatic disease, or has recurred during, or within 6 months of completing, an irinotecan-containing adjuvant regimen, or other histologically-confirmed solid tumors refractory to standard therapy.
* Age at least 18 years at the time of the first dose of study drug.
* Both males and females are eligible. Sexually active females, unless surgically sterile (or at least one year post-menopausal), must have used an effective method of avoiding pregnancy (including oral or implanted contraceptives, IUD, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 30 days prior to the first dose of study drug, and must agree to continue using such precautions for 30 days after the final dose of study drug. Sexually active females of reproductive potential must have a negative serum b human chorionic gonadotropin (bhCG) pregnancy test within 3 days of start of therapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. ECOG criteria are described in Appendix A.
* Patients who had prior treatment with chemotherapy or radiotherapy or had prior surgery are eligible for study entry if at least 4 weeks have past since their treatment/surgery.
* All toxicities related to prior treatment must have resolved and all surgical wounds must have healed.
* Prior immunotherapy with approved agents is allowable.
* ANC ³1500/mm3, platelets ³100,000/mm3, hemoglobin >10.0 g/dL, serum creatinine £1.5 mg/dL or calculated creatinine clearance >50 mL/min, serum bilirubin £2.0 mg/dL, and AST/ALT £5 times the upper limit of normal (ULN).
* PT/PTT less than ULN or international normalized ratio (INR) less than 1.12.
* Thyroxine (T4) and thyroid-stimulating hormone (TSH) within normal limits.
* Written informed consent obtained from the patient prior to receipt of any study medication or beginning study procedures.

Exclusion Criteria:

* Pregnancy or nursing.
* Known brain metastases or primary brain tumors, symptomatic pleural effusion or ascites requiring paracentesis.
* Respiratory insufficiency requiring oxygen treatment, or lymphangitic involvement of lungs.
* Any evidence of hematemesis, melena, hematochezia, or gross hematuria.
* A history of significant adverse events related to a previously administered humanized monoclonal antibody.
* A known human immunodeficiency virus (HIV) or hepatitis virus infection.
* A prior myocardial infarction or angina, or uncontrolled hypertension (systolic blood pressure >150 mm Hg).
* A prior stroke or transient ischemic attack.
* An active infection requiring systemic antiinfective therapy.
* Received an investigational agent in the last 4 weeks of initiation of study treatment.
* A requirement for palliative chemotherapy, hormonal therapy, or immunotherapy during the course of the study.
* Clinical evidence of bowel obstruction.
* A history of other malignancies within the past 5 years (with the exception of basal cell carcinoma of the skin or completely excised in situ carcinoma of the cervix).
* A general medical or psychological condition or behavior, including substance dependence or abuse that, in the opinion of the investigator, might not permit the patient to complete the study or sign the informed consent.
* Prior treatment with MEDI-522 or MEDI-523.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2001-07; Primary Completion 2005-01 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
The recommended Phase II dose will be based on acceptable dose-limiting toxicity | Study Days 0, 7, 14, 21, 28, 35, 42, and 49.

SECONDARY OUTCOMES:
Pharmacokinetic parameters may also be factored into the determination of a Phase II dose and; Tumor response | Study Days 0, 28, 56, 84, 112, 140, 168, 196, 224, 252, 280, 308, 336, 357; and tumor response on Study Days 56, 112, 168, 224, 280, 336, and 387.

CONTACTS AND LOCATIONS:
Overall Officials: Krista Arbaugh, Dir., Clinical Ops, Study Director — MedImmune LLC
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States